CLINICAL TRIAL: NCT02999230
Title: Probiotics That Moderate pH and Antagonize Pathogens to Promote Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB201602471-N; 5R01DE025832-05 (NIH)
Record Dates: First submitted 2016-12-13; First posted 2016-12-21 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
Keywords: Cavities
MeSH Terms: conditions — Dental Caries | interventions — Arginine; Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Caries Free (Active Comparator): Gums will be examined and caries assessment performed. On some visits Saliva and supragingival plaque will be collected. Study toothpaste will be assigned.
  Interventions: Other: Caries Free 1.5% Arginine
- Caries Free- Placebo (Placebo Comparator): Gums will be examined and caries assessment performed. On some visits Saliva and supragingival plaque will be collected. Marketed Toothpaste will be assigned.
  Interventions: Other: Caries Free Placebo Sodium Fluoride
- Caries Active (Active Comparator): Gums will be examined and caries assessment performed. On some visits Saliva and plaque will be collected. Study toothpaste will be assigned.
  Interventions: Other: Caries Active 1.5% Arginine
- Caries Active- Placebo (Placebo Comparator): Gums will be examined and caries assessment performed. On some visits Saliva and supragingival plaque will be collected. Marketed Toothpaste will be assigned.
  Interventions: Other: Caries Active- Placebo Sodium Fluoride

INTERVENTIONS:
Other: Caries Free 1.5% Arginine — Study toothpaste assigned containing 1.5% Arginine. Subjects will also receive a Colgate Wave Comfort Adult Toothbrush to brush their teeth with twice a day.
  Other Names: 1.5% Arginine
  Arms: Caries Free
Other: Caries Free Placebo Sodium Fluoride — Marketed Toothpaste containing 1100 ppm F as Sodium Fluoride will be assigned. Subjects will also receive a Colgate Wave Comfort Adult Toothbrush to brush their teeth with twice a day.
  Other Names: Sodium Fluoride
  Arms: Caries Free- Placebo
Other: Caries Active 1.5% Arginine — Study toothpaste assigned containing 1.5% Arginine. Subjects will also receive a Colgate Wave Comfort Adult Toothbrush to brush their teeth with twice a day.
  Other Names: 1.5% Arginine
  Arms: Caries Active
Other: Caries Active- Placebo Sodium Fluoride — Marketed Toothpaste containing 1100 ppm F as Sodium Fluoride will be assigned. Subjects will also receive a Colgate Wave Comfort Adult Toothbrush to brush their teeth with twice a day.
  Other Names: Sodium Fluoride
  Arms: Caries Active- Placebo

SUMMARY:
This study will examine the mechanisms of action of probiotics and synbiotics for control of oral diseases, with a particular focus on exploring new strategies for caries prevention and treatment.

DETAILED DESCRIPTION:
Subjects recruited in years 1, 2, and 4 will only be seen for one study visit and will follow the research visit protocol listed below:

Pre-Screening - If the subject chooses to be pre-screened for this study they will be asked to fill out a study registration form and an oral habits/medical history form. They will be asked to sign an Informed Consent. The subject will then have their teeth and gums examined. At this visit, the investigator will assess whether or not the subject is a good candidate for the study. During the phone interview each subject was asked not to brush or floss their teeth and not to eat or drink anything other than water for 8 hours prior to the pre-screening visit (Visit 0). If the subject was compliant with these requests, oral samples will be collected at this pre-screening visit and will now be considered Visit 1 (Baseline). If not, they will be asked to return to the clinic for another visit and asked not to brush or floss their teeth and not to eat or drink anything other than water 8 hours prior to that appointment. This visit will then be consider Visit 1 (Baseline).

Visit 1 (Baseline) - The subject will have their medical and dental history reviewed. They will have their teeth and gums examined. Saliva and plaque will be collected. This will be the end of the study for subjects recruited in years 1, 2, and 4.

Subjects will be grouped by the year they participate in the study. Subjects recruited in year 3 will follow the research visit protocol outlined below:

Pre-Screening - If the subject chooses to be pre-screened for this study they will be asked to fill out a study registration form and an oral habits/medical history form. They will be asked to sign an Informed Consent. The subject will then have their teeth and gums examined. At this visit, the investigator will assess whether or not the subject is a good candidate for the study. During the phone interview each subject was asked not to brush or floss their teeth and not to eat or drink anything other than water for 8 hours prior to the pre-screening visit (Visit 0). If the subject was compliant with these requests, oral samples will be collected at this pre-screening visit and will now be considered Visit 1 (Baseline). If not, they will be asked to return to the clinic for another visit and asked not to brush or floss their teeth and not to eat or drink anything other than water 8 hours prior to that appointment. This visit will then be considered Visit 1 (Baseline).

Visit 1 (Baseline) - The subject will have their medical and dental history reviewed. They will have their teeth and gums examined. Saliva and plaque will be collected. Each subject will be given a toothbrush and toothpaste and instructed to not use any other dental products. This will be considered the "washout" period.

Visit 2 - The subject will be asked to return the unused toothpaste. Their medical and dental history will be reviewed and they will have their teeth examined. Saliva and plaque will be collected at this visit. The subjects will then be randomly assigned (by chance, like the flip of a coin) to the group that will use a marketed fluoride-containing toothpaste or to the group that will use a marketed arginine containing toothpaste. The subject will also be instructed not to brush or floss their teeth or eat or drink anything other than water for 8 hours prior to the next appointment.

Visits 3, 4, and 5 - Subjects will not be allowed to brush or floss their teeth or eat or drink anything other than water 8 hours prior to these visits. Saliva and plaque will be collected. On the 5th visit subjects will be asked to return the unused toothpaste tube. At this time participation in this research study will end and they will be instructed to return to their regular oral hygiene regiments.

ELIGIBILITY:
Inclusion Criteria:

* Twenty natural uncrowned teeth excluding third molars
* No contraindications to dental treatment
* Caries Free-(with no clinical evidence of past or present caries)
* Caries Active- (At least two active sites)

Exclusion Criteria:

* Less than 20 teeth
* Systemic disease that can cause xerostomia
* Taking medication known to cause xerostomia
* Have been treated with antibiotics within the past 3 months
* Advanced periodontal disease
* Removable or fixed dental appliances
* Bleeding disorders or taking anticoagulant medications
* Immune compromised individuals
* Uses tobacco products
* Participation in another clinical study one week prior to the start of the washout period or during the study period
* Use of any flavored products, such as mint flavored candies and chewing gum, one week prior to or during the study
* Unwilling or unable to provide informed consent and follow plaque/saliva collection instructions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from baseline to week 2 | Changes from baseline to 2 weeks (Screening)
  Saliva and dental plaque will be collected during the baseline and week 2 study visits. The amount of ammonia and/or citrulline produced via the ADS by oral bacteria present in the collected oral samples will be measured and compared using standardized protocols.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from week 2 to week 4 | Changes from week 2 to week 4 (Baseline)
  Saliva and dental plaque will be collected during the week 2 and week 4 study visits. The amount of citrulline and/or ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured and compared using standardized protocols.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from week 4 to week 8 | Changes from week 4 to week 8 (Washout)
  Saliva and dental plaque will be collected during the week 4 and week 8 study visits. The amount of ammonia and/or citrulline produced via the ADS by oral bacteria present in the collected oral samples will be measured and compared using standardized protocols.
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from week 8 to week 12 | Changes from week 8 to week 12 (Evaluation)
  Saliva and dental plaque will be collected during the week 8 and week 12 visits. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured and compared using standardized protocols
Levels of the arginine deiminase system (ADS) in oral samples of healthy and caries-active subjects changes from baseline to week 12. | Changes from baseline to week 12 (Evaluation)
  Saliva and dental plaque will be collected during the baseline and week 12 study visits. The amount of ammonia produced via the ADS by oral bacteria present in the collected oral samples will be measured and compared using standardized protocols.

SECONDARY OUTCOMES:
Bacteria collected from oral samples of healthy and caries-active subjects changes from baseline to week 2 | Changes from baseline to week 2
  Saliva and dental plaque will be collected during the baseline and week 2 study visits.Bacteria present in these oral samples will be isolated and identified. The capacity of the bacteria to produce ammonia from arginine in different environmental conditions will be measured.
Bacteria collected from oral samples of healthy and caries-active subjects changes from week 2 to week 4 | Changes from week 2 to week 4
  Saliva and dental plaque will be collected during the week 2 and week 4 study visits. Bacteria present in these oral samples will be isolated and identified. The capacity of the bacteria to produce ammonia from arginine in different environmental conditions will be measured.
Bacteria collected from oral samples of healthy and caries-active subjects changes from week 4 to week 8 | Changes from week 4 to week 8
  Saliva and dental plaque will be collected during the week 4 to week 8 study visits. Bacteria present in these oral samples will be isolated and identified. The capacity of the bacteria to produce ammonia from arginine in different environmental conditions will be measured.
Bacteria collected from oral samples of healthy and caries-active subjects changes from week 8 to week 12 | Changes from week 8 to week 12
  Saliva and dental plaque will be collected during the week 8 and week 12 study visits. Bacteria present in these oral samples will be isolated and identified. The capacity of the bacteria to produce ammonia from arginine in different environmental conditions will be measured.
Bacteria collected from oral samples of healthy and caries-active subjects changes from baseline to week 12 | Changes from baseline to week 12
  Saliva and dental plaque will be collected during the baseline and week 12 study visits. Bacteria present in these oral samples will be isolated and identified. The capacity of the bacteria to produce ammonia from arginine in different environmental conditions will be measured.

OTHER OUTCOMES:
Salivary factors present in healthy and caries-active subjects during the research study. | Up to 6 months
  Saliva will be collected from healthy and caries-active subjects during the research study. The differences in salivary factors between the healthy and caries-active groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle Nascimento, DDS, MS PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Dentistry, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No